CLINICAL TRIAL: NCT04533971
Title: The Effect of a Series of Systemic Cryotherapy Treatments on the Bioelectrical Activity of Muscles and the Functional State of Patients With Multiple Sclerosis
Brief Title: The Effect of a Series of Systemic Cryotherapy Treatments on the Functional State of Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Anna Lubkowska, Profesor, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2016.01.01
Record Dates: First submitted 2020-08-18; First posted 2020-09-01 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2020-08

CONDITIONS: Multiple Sclerosis (ICD10-G35)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to the two groups, WBC and control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WBC group (Experimental): Criteria
  * documented diagnosis of MS,
  * functional status classified according to the Expanded Disability Status Scale (EDSS) to a level lower or equal to 0-3
  * no contraindications for WBC treatments found in the medical examination
  * no other serious chronic diseases identified that may affect the results of the tests carried out
  * readiness to participate in daily WBC
  * a written statement of volunteers about not using WBC treatments in the last 2 years, and not using other forms of physiotherapeutic and complementary therapies (other than planned in the procedures) for the period of this study
  Interventions: Other: Whole body cryotherapy
- Control Group (No Intervention): Criteria
  * documented diagnosis of MS,
  * functional status classified according to the Expanded Disability Status Scale (EDSS) to a level lower or equal to 0-3
  * no contraindications for WBC treatments found in the medical examination
  * no other serious chronic diseases identified that may affect the results of the tests carried out
  * readiness to participate in daily WBC
  * a written statement of volunteers about not using WBC treatments in the last 2 years, and not using other forms of physiotherapeutic and complementary therapies (other than planned in the procedures) for the period of this study

INTERVENTIONS:
Other: Whole body cryotherapy — The WBC procedure consisted of 2-3 min walk in the cryogenic chamber at -110℃. Immediately before the WBC procedures, the patients were provided with a special treatment suit, they were instructed as to how to protect the parts of the body that are particularly vulnerable to frostbite, on the proper way of moving and breathing during the treatment. Excluding Saturdays and Sundays, the WBC treatments were performed daily for the next four weeks. Each time after the WBC the subjects participated in 15-minute kinesitherapy exercises conducted in groups of 5-6 people. The exercises were of general improvement nature and took into account the mobility of the subjects.
  Arms: WBC group

SUMMARY:
Multiple sclerosis (Latin: Sclerosis multiplex; MS) is a chronic, inflammatory and degenerative disease of the central nervous system (CNS) characterised by a varied course and symptomatology. The chronic nature of the disease and gradual loss of tissue within the CNS result in increasing neurological deficits and motor failure over time. Due to the characteristics of the symptoms and the chronic course of MS, patients with MS use various forms of physiotherapeutic procedures throughout most of their lives, including especially often whole-body cryotherapy (WBC) treatments. The aim of this study was to assess potential changes in bioelectrical muscle activity during rest and contraction after exposure on 20 series of Whole body cryotherapy (WBC) in patients with multiple sclerosis (MS). Assessment potential relationships between the sEMG parameters and functional state in patients with multiple sclerosis pre and post 20 series of WBC.

Finally, 114 patients with MS participated in the planned procedures of research. The participants were randomly assigned to the two groups, WBC and control. The sample size was 60 in WBC, and 54 in control groups. Testing before and after series of WBC consisted of: clinical assessment of fatigue was performed by the Fatigue Severity Scale (FSS), gait speed using Timed 25 Foot Walk (T25-FW), Hand grip strength (HGS), and surface electromyography (sEMG) of the dominant hand.

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of MS,
* functional status classified according to the Expanded Disability Status Scale (EDSS) to a level lower or equal to 0-3
* no contraindications for WBC treatments found in the medical examination
* no other serious chronic diseases identified that may affect the results of the tests carried out
* readiness to participate in daily WBC
* a written statement of volunteers about not using WBC treatments in the last 2 years, and not using other forms of physiotherapeutic and complementary therapies (other than planned in the procedures) for the period of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2015-04-01; Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Assessment of changes in the level of fatigue | On the day preceding the start of a 20 series of WBC ( 4 weeks) ( T0) and between the second and the fourth day, after the end of a series of WBC (T1).
  The assessment tool: Fatigue Severity Scale (FSS). The FSS questionnaire is composed of 9 items related to the severity of symptoms commonly present in MS patients. Each question is rated on a scale of 1 to 7 (where 1 - "strongly disagree", 7 - "strongly agree").
  Minimum value: 9 points (if you answer "1" to all questions) Maximum value: 63 points (if you answer "7" to all questions) A higher score indicates greater fatigue intensity - i.e. a worse result. A score of ≥ 36 points is considered significantly elevated and indicates significant fatigue intensity.
Assessment of changes in walking speed | On the day preceding the start of a 20 series of WBC ( 4 weeks) ( T0) and between the second and the fourth day, after the end of a series of WBC (T1).
  The aassessment tool: 25 Foot Walk (T25-FW) Maximal walking speed, across a clearly marked, linear 25-foot (7.62-m course). The T25-FW score was an average in seconds from the two successive trials
Assessment of changes in hand grip strength | On the day preceding the start of a 20 series of WBC ( 4 weeks) ( T0) and between the second and the fourth day, after the end of a series of WBC (T1).
  The aassessment tool: hand grip strength (HGS). Dominant hand. HGS measurements were performed in according to the recommendations of the American Society of Hand Therapists
Assessment of changes in the bioelectrical activity of muscles. | On the day preceding the start of a 20 series of WBC ( 4 weeks) ( T0) and between the second and the fourth day, after the end of a series of WBC (T1).
  The aassessment tool: surface electromyography (sEMG) of the dominant hand. The sEMG test was performed for extensor (ECR - Extensor carpi radialis) and a flexor (FCR- Flexor carpi radialis) muscles of the wrist, for the dominant hand.
  * 30-second electromyographic signal in the resting position
  * 2 isometric maximal voluntary contractions (MVC) of five seconds against a fixed handle separated by 90 s rest, for FCR and ECR of the dominant side.
  * voluntary contraction during 10 sec (wrist flexion and next extension against the fixed plates). Recording of VC repeated three times.

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Radecka, Principal Investigator — Department of Functional Diagnostics and Physical Medicine, PUM; Anna Lubkowska, Profesor, Study Director — Department of Functional Diagnostics and Physical Medicine, PUM; Anna Knyszyńska, PhD, Study Chair — Department of Functional Diagnostics and Physical Medicine, PUM

IPD SHARING:
Plan to Share IPD: No